CLINICAL TRIAL: NCT05639946
Title: Brivaracetam to Reduce Neuropathic Pain in Chronic SCI: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PMR-2022-30886
Record Dates: First submitted 2022-11-23; First posted 2022-12-07 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries; Neuropathic Pain
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia | interventions — brivaracetam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants with severe neuropathic pain will receive brivaracetam treatment
  Interventions: Drug: brivaracetam
- Control group (Placebo Comparator): Participants with severe neuropathic pain will receive placebo drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: brivaracetam — Drug dosage will be individually titrated for each participant with a goal of 100mg BID according to the following dose escalation protocol that we use clinically: 50mg BID for 2 weeks, followed by 50mg TID for 2 weeks, followed by 100mg BID for 48 days as tolerated. Participants will be allowed to reduce the dose of brivaracetam if they experience unacceptable side effects defined as increased somnolence according to routine clinical practice with other drugs in this class used for pain.
  Arms: Experimental group
Drug: Placebo — Participants will receive placebo drug
  Arms: Control group

SUMMARY:
Spinal cord injury (SCI) is associated with severe neuropathic pain that is often refractory to pharmacological intervention. Preliminary data suggest brivaracetam is a mechanism-based pharmacological intervention for neuropathic pain in SCI. Based on this and other reports in the literature, SCI-related neuropathic pain is hypothesized to occur largely because of upregulation of synaptic vesicle protein 2A (SV2A) within the substantia gelatinosa of the injured spinal cord. Furthermore, compared to placebo, brivaracetam treatment is hypothesized to reduce severe below-level SCI neuropathic pain and increases parietal operculum (partsOP1/OP4) connectivity strength measured by resting-state functional Magnetic Resonance Imaging (rsfMRI). Circulating miRNA-485 levels may be associated with change in pain intensity due to brivaracetam treatment. The study aims to determine the efficacy of brivaracetam treatment for SCI-related neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Injured for > 3 months
* Completed inpatient rehabilitation and living in the community
* Chronic sublesional neuropathic pain defined as persistent pain (VAS grade 3-10) for three months or more
* For people of child-bearing potential: currently practicing an effective form of two types of birth control (defined as those, alone or in combination, that result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly).

Exclusion Criteria:

* Progressive myelopathy secondary to posttraumatic cord tethering or syringomyelia
* Active use of drugs known to interact with brivaracetam: rifampin, carbamazepine, sodium oxybate, buprenorphine, propoxyphene, levetiracetam, and phenytoin.
* Brain injury or cognitive impairment limiting the ability to follow directions or provide informed consent
* Pregnancy or lactation
* Epilepsy or active treatment for seizure disorder
* Past or current suicidality
* Active treatment for psychiatric disease
* Drug addiction
* Moderate or heavy alcohol intake (up to four alcoholic drinks for men and three for women in any single day, and a maximum of 14 drinks for men and 7 drinks for women per week)
* Hepatic cirrhosis, Child-Pugh grades A, B, and C
* Impaired renal function (GFR<60ml/minute)
* Contraindications to brivaracetam or pyrrolidine derivatives including allergy
* Active clinically significant disease (e.g., renal, hepatic, neurological, cardiovascular, pulmonary, endocrine, psychiatric, hematologic, urologic, or other acute or chronic illness) that, in the opinion of the investigator, would make the patient an unsuitable candidate for this trial.
* History of malabsorption or other gastrointestinal (GI) disease that may significantly alter the absorption of brivaracetam
* Use of any investigational drug 30 days prior to enrollment in this study
* Enrollment in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
change in pain intensity | 3 months
  the International Spinal Cord Injury Pain Data Set
change in operculum brain connectivity | 3 months
  assess changes in cortical activity of related pain perception regions and networks in the brain in response to brivaracetam treatment compared to placebo using rsfMRI and pain- related task-based fMRI.
microRNA-485 levels | baseline
  use Next-Generation sequencing to assess miR-485 levels
microRNA-485 levels | 3 months
  use Next-Generation sequencing to assess miR-485 levels

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Battaglino, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States